CLINICAL TRIAL: NCT05167734
Title: The Practical Anemia Bundle for SusTained Blood Recovery (PABST-BR) Clinical Trial
Brief Title: Practical Anemia Bundle for SusTained Blood Recovery
Acronym: PABST-BR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Matthew A. Warner, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-006511; K23HL153310-01 (NIH)
Record Dates: First submitted 2021-11-30; First posted 2021-12-22 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Anemia; Critical Illness
MeSH Terms: conditions — Anemia; Critical Illness | interventions — Iron-Dextran Complex; Erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Standard of Care) Group (No Intervention): Subjects will receive standard clinical care for the treatment of anemia while in the ICU.
- Anemia Treatment Bundle (Experimental): The intervention arm is multi-faceted with 3 primary components: 1) Optimized phlebotomy, defined by minimal volume draws and closed-loop blood sampling, all performed by a dedicated phlebotomy team independent from the treatment team; 2) Decision support aids, including visual and electronic alerts reminding the care team to minimize non-essential laboratory testing and mitigate patient-specific bleeding risk; and 3) Pharmacologic anemia treatment with a single dose of IV iron and/or subcutaneous erythropoietin (given immediately following enrollment) targeted to 2 broad groups: 1) anemias responsive to iron supplementation alone (i.e. acute blood loss, iron deficiency) and 2) anemias requiring erythropoietic stimulation (e.g. anemia of inflammation, anemia of renal disease).
  Interventions: Drug: Iron Dextran; Drug: Erythropoietin (EPO)

INTERVENTIONS:
Drug: Iron Dextran — 1000 mg IV
  Arms: Anemia Treatment Bundle
Drug: Erythropoietin (EPO) — 40,000 units subcutaneous
  Other Names: EPO
  Arms: Anemia Treatment Bundle

SUMMARY:
The purpose of this study is to test a multi-faceted anemia treatment plan to reduce the severity of anemia and to promote hemoglobin and functional recovery in adults who have been in the intensive care unit (ICU).

DETAILED DESCRIPTION:
Anemia is common during critical illness and is associated with impaired outcomes during and after hospitalization. The goal of this investigation is to test a multi-faceted anemia prevention and targeted treatment bundle to attenuate anemia development and promote functional recovery in the setting of critical illness. Specifically, this will be a pragmatic phase II clinical trial of a multi-faceted anemia prevention and treatment bundle with 3 aspects (optimized phlebotomy practice, clinical decision support, targeted pharmacologic anemia treatment) assessing the impact of the intervention on hemoglobin concentrations (primary aim), transfusion utilization, and functional outcomes through 3 months after hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form (may be completed by legal proxies for those patients unable to provide consent, i.e. sedation/intubation)
* Stated willingness to comply with all study procedures and availability for the duration of the study, including follow-up assessments
* Current ICU admission at Mayo Clinic Rochester with anticipated ICU duration >48 hours after enrollment
* Current ICU duration < 7 days
* Patients embedded in the local or regional Mayo Clinic Health System to facilitate post-hospitalization outcome assessment
* Moderate-to-severe anemia (i.e. hemoglobin concentration < 10 g/dL) at the time of enrollment, with the hemoglobin concentration assessed no more than 24 hours prior to enrollment. If RBC transfusion has been administered between the qualifying hemoglobin assessment and enrollment, a repeat hemoglobin will be required prior to enrollment to ensure that it remains < 10 g/dL.

Exclusion Criteria:

* Recent or current IV iron or erythropoiesis stimulating agent (ESA) use (i.e. darbepoetin, Aranesp, erythropoietin, Epogen, Procrit, Retacrit) within 30 days of enrollment
* Severe anemia prior to hospitalization (i.e. hemoglobin <9 g/dL within 90 days of admission)
* Known allergic reactions to iron or EPO
* Inability to complete outcome assessments (i.e. not expected to survive hospitalization, unable to make follow-up appointments, non-ambulatory, dementia or other severe cognitive impairment, visual impairment i.e. blind or legally blind)
* Pregnancy or breastfeeding at time of enrollment
* Inability to receive pharmacologic venous thromboembolic prophylaxis except in patients with recent surgical or gastrointestinal bleeding
* Active or suspected thrombosis (i.e. deep venous thrombosis, pulmonary embolism, acute arterial thrombus within 3 months)
* Uncontrolled sepsis (i.e. <48 hours of appropriate antimicrobial therapy and/or lack of definitive source control)
* Having received ≥10 units of allogeneic RBCs in the 48 hours before enrollment
* Acute coronary syndrome or ischemic stroke within 3 months
* Weight less than 40 kg
* Concerns with study enrollment expressed by the clinical team
* Mechanical circulatory support devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Warner, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Study data will be shared through the NHLBI Data Repository, which is managed by thenBiologic Specimen and Data Repository Information Coordinating Center (BioLINCC). In addition to study data (e.g. information recorded for each study participant including demographics, clinical characteristics, laboratory assessments, and outcomes / follow-up assessments), study documentation information will also be provided in order to facilitate secondary use of data by investigators not familiar with the original data set. This includes a summary documentation file, manuals of procedures, detailed statistical code, and data dictionary information, among other important documentation. The timing and manner of research data uploading to the Data Repository will be in full compliance with NHLBI guidelines.
Time Frame: We commit to providing data immediately upon acceptance of the data for scientific publication or within one year of completion of the award period (whichever comes first).
Access Criteria: All published scientific manuscripts will contain information regarding how to request and access study data.

REFERENCES:
- [Derived] Warner MA, Johnson ML, Hanson AC, Fortune E, Flaby GW, Schulte PJ, Hazelton VM, Go RS, Beam WB, Charnin JE, Anderson BK, Karon B, Cheville AL, Gajic O, Kor DJ. Practical Anemia Bundle and Hemoglobin Recovery in Critical Illness: A Randomized Clinical Trial. JAMA Netw Open. 2025 Mar 3;8(3):e252353. doi: 10.1001/jamanetworkopen.2025.2353. PMID 40152861
- [Derived] Warner MA, Go RS, Schulte PJ, Beam WB, Charnin JE, Meade L, Droege KA, Anderson BK, Johnson ML, Karon B, Cheville A, Gajic O, Kor DJ. Practical Anemia Bundle for Sustained Blood Recovery (PABST-BR) in critical illness: a protocol for a randomised controlled trial. BMJ Open. 2022 Dec 2;12(12):e064017. doi: 10.1136/bmjopen-2022-064017. PMID 36460332

RESULTS

PARTICIPANT FLOW:
Groups:
- Control (Standard of Care) Group: Subjects received standard clinical care for the treatment of anemia while in the ICU.
Period: Overall Study
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Started | 51 | 49
Completed | 51 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (11.6) | 65.4 (9.3) | 65.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 43
  Male | 28 | 29 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 50 | 48 | 98
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 48 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 51 | 49 | 100

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Concentrations
Description: Hemoglobin is a protein that cares oxygen through the body
Time Frame: 1 month post-hospitalization
Population: Data was not collected nor analyzed for four subjects in the Control (Standard of Care) Group and eight subjects in the Anemia Treatment Bundle arm
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 47 | 41
g/dL | 11.5 [10.3 to 12.6] | 12.2 [11.8 to 13.0]
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; Test type: Superiority; p = 0.02, Mixed Models Analysis; linear mixed effects model adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Mean Difference (Final Values) = 0.7, 95% CI 2-sided [0.1 to 1.2] — values greater than 0 infer higher hemoglobin in active intervention

2. Secondary Outcome: Hemoglobin Concentrations
Description: Hemoglobin is a protein that cares oxygen through the body
Time Frame: Hospital discharge (approximately 1 month), 3 months post-hospitalization
Population: Data was not collected or analyzed for 8 subjects in the control standard of care arm and 7 subjects in the anemia treatment bundle arm at 3-months post hospitalization.
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 51 | 49
g/dL
  Hospital discharge | 9.0 [8.6 to 10.0] | 9.6 [8.9 to 9.9]
  3-months post hospitalization: number analyzed (Participants) | 43 | 42
  3-months post hospitalization | 12.8 [11.7 to 13.8] | 13.4 [12.2 to 14.6]
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 3-months post hospitalization; Test type: Superiority; p = 0.04, Mixed Models Analysis; linear mixed effects model adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [0.0 to 1.1] — adjusted mean difference
Statistical Analysis 2: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; Hospital Discharge; Test type: Superiority; p = 0.42, Mixed Models Analysis; linear mixed effects model adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.3 to 0.7]

3. Secondary Outcome: Phlebotomy Practice-Blood Draws
Description: Number of times subjects have blood drawn
Time Frame: Hospital discharge (approximately 1 month)
Measure: Median (Inter-Quartile Range); unit: Number of blood draws
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 51 | 49
Number of blood draws | 46 [20 to 74] | 32 [24 to 55]
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; Test type: Superiority; p = 0.352, Mixed Models Analysis

4. Secondary Outcome: Phlebotomy Practice-Volume
Description: Total volume of phlebotomy blood draws
Time Frame: Hospital discharge (approximately 1 month)
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 51 | 49
mL | 142 [68 to 195] | 32 [22 to 54]
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; Test type: Superiority; p < 0.001, Mixed Models Analysis — threshold for significance - p<0.05

5. Secondary Outcome: Patient-Reported Quality of Life Measured by EuroQol (EQ-5D)
Description: The EuroQol (EQ-5D) is a 5-item questionnaire that assess health-related quality of life over five different dimensions of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Total score ranges from 0 to 100, with higher scores indicating improved health.
Time Frame: Hospital discharge (approximately 1 month), 1 month post-hospitalization, 3 months post-hospitalization
Population: Data was not collected nor analyzed for 1 subject in the Control (Standard of Care) arm and 1 subject in the Anemia Treatment Bundle arm at hospital discharge. No data was collected or analyzed for 6 subjects in the control standard of care arm and 7 subjects in the anemia treatment bundle arm at 1-month post hospitalization. No data was collected or analyzed for 10 subjects in the control standard of care arm and 8 subjects in the anemia treatment bundle arm at 3-months post hospitalization.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 50 | 48
score on a scale
  Hospital discharge | 60 [40 to 70] | 51 [40 to 75]
  1 month post hospitalization: number analyzed (Participants) | 45 | 42
  1 month post hospitalization | 65 [50 to 75] | 70 [65 to 80]
  3 months post hospitalization: number analyzed (Participants) | 41 | 41
  3 months post hospitalization | 80 [75 to 85] | 80 [75 to 90]
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; Hospital Discharge; Test type: Superiority; p = 0.94, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.44 to 2.40] — Estimates are odds ratios and correspond to the multiplicative increase in odds of higher value/score associated with active intervention
Statistical Analysis 2: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 1-month post hospitalization; Test type: Superiority; p = 0.18, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 1.79, 95% CI 2-sided [0.76 to 4.20] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 3-months post hospitalization; Test type: Superiority; p = 0.64, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.51 to 3.00] — [estimate comment as in outcome 5, analysis 1]

6. Secondary Outcome: Anemia-related Fatigue Measured by Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale is a 13-item questionnaire used to measure the severity of fatigue and its impact on daily activities. Each question is rated on a 4-point scale where 0 represents "very much" fatigued and 4 represents "not at all" fatigued. Total scores range from 0 to 52 with lower scores indicating greater fatigue.
Time Frame: Hospital discharge (approximately 1 month), 1 month post-hospitalization, 3 months post-hospitalization
Population: Data was not collected or analyzed for 1 subject in the Control Standard of Care arm and 1 subject in the Anemia Treatment Bundle arm at hospital discharge. No data was collected or analyzed for 6 subjects in the control standard of care arm and 7 subjects in the anemia treatment bundle arm at the 1-month post hospitalization. No data was collected or analyzed for 10 subject in the control standard of care arm and 8 subject in the anemia treatment bundle arm at the 3-months post hospitalization.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 50 | 48
score on a scale
  Hosptial Discharge | 28 [19 to 36] | 32 [24 to 37]
  1 month post hospitalization: number analyzed (Participants) | 45 | 42
  1 month post hospitalization | 37 [25 to 43] | 41 [32 to 45]
  3 months post hospitalization: number analyzed (Participants) | 41 | 41
  3 months post hospitalization | 44 [40 to 46] | 46 [41 to 48]
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; Hospital discharge; Test type: Superiority; p = 0.23, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 1.81, 95% CI 2-sided [0.68 to 4.80] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 1-month post hospitalization; Test type: Superiority; p = 0.09, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 2.43, 95% CI 2-sided [0.87 to 6.80] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 3-months post hospitalization; Test type: Superiority; p = 0.084, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 2.52, 95% CI 2-sided [0.88 to 7.20] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: 6 Minute Walk Distance
Description: Distance walked in 6 minutes used to assess physical function after critical illness.
Time Frame: 1 and 3-months post-hospitalization
Population: No data was collected or analyzed for 33 participants in the control standard of care arm and 32 participants in the anemia treatment bundle arm at 1-month post hospitalization. No data was collected or analyzed for 39 participants in the control standard of care arm and 41 participants in the anemia treatment bundle arm at 3-months post hospitalization.
Measure: Median (Inter-Quartile Range); unit: Feet
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 18 | 17
Feet
  1 month post hospitalization | 1080 [790 to 1250] | 1211 [960 to 1480]
  3 months post hospitalization: number analyzed (Participants) | 12 | 8
  3 months post hospitalization | 1208 [880 to 1733] | 1220 [1040 to 1683]
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 1-month post hospitalization; Test type: Superiority; p = 0.13, Mixed Models Analysis; adjusting for baseline hemoglobin, age, sex, surgical vs. non-surgical admission, and baseline ADLs; Mean Difference (Net) = 218, 95% CI 2-sided [-73 to 510] — scores greater than 0 reflect greater ambulatory distance in active intervention
Statistical Analysis 2: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 3-months post hospitalization; Test type: Superiority; p = 0.27, Mixed Models Analysis; adjusting for baseline hemoglobin, age, sex, surgical vs. non-surgical admission, baseline ADLs; Median Difference (Net) = 178, 95% CI 2-sided [-154 to 510]

8. Secondary Outcome: Cognitive Function After Critical Illness Assessed Using Montreal Cognitive Assessment (MoCA-BLIND)
Description: The Montreal Cognitive Assessment (MoCA-BLIND) score assesses cognitive impairment by a 30-item questionnaire that includes tests of orientation, attention, memory, language and visual-spatial skills. Possible scores range from 0 to 30, with higher scores indicating higher cognitive function. A final total score of 26 and above is considered normal.
Time Frame: 1 and 3-months post-hospitalization
Population: No data was collected or analyzed for 11 participants in the control standard of care arm and 10 participants in the anemia treatment bundle arm at 1-month post hospitalization. No data was collected or analyzed for 14 participants in the control standard of care arm and 13 participants in the in the anemia treatment bundle arm at 3-months post hospitalization.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 40 | 39
score on a scale
  1 month post hospitalization | 19 [18 to 21] | 20 [19 to 22]
  3 months post hospitalization: number analyzed (Participants) | 37 | 36
  3 months post hospitalization | 20 [20 to 21] | 21 [20 to 22]
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 1-month post hospitalization; Test type: Superiority; p = 0.12, proportional odds; adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 2.49, 95% CI 2-sided [0.79 to 7.80] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 3-months post hospitalization; Test type: Superiority; p = 0.07, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 3.10, 95% CI 2-sided [0.91 to 10.5] — [estimate comment as in outcome 5, analysis 1]

9. Secondary Outcome: Mental Health - Anxiety and Depression Measured Using the Hosptial Anxiety and Depression Scale (HADS)
Description: The Hospital Anxiety and Depression Scale (HADS) assesses a patient's anxiety and depression levels. Subject's answer 14 questions (7 for anxiety and 7 for depression). Each question is scored from 0-3. Total scores can range from 0 to 21 for either anxiety or depression, with higher scores indicating a presence of anxiety or depression.
Time Frame: 1 and 3-months post-hospitalization
Population: No data was collected or analyzed for 6 participants in the control standard of care arm and 7 participants in the anemia treatment bundle arm at 1-month post hospitalization. No data was collected or analyzed for 10 participants in the control standard of care arm and 8 in the anemia treatment bundle arm at 3-months post hospitalization.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 45 | 42
score on a scale
  Anxiety Score-1 month post hospitalization | 2 [1 to 3] | 1 [0 to 3]
  Anxiety Score-3 months post hospitalization: number analyzed (Participants) | 41 | 41
  Anxiety Score-3 months post hospitalization | 1 [0 to 3] | 0 [0 to 5]
  Depression Score-1 month post hospitalization | 4 [1 to 7] | 2 [1 to 5]
  Depression Score-3 months post hospitalization: number analyzed (Participants) | 41 | 41
  Depression Score-3 months post hospitalization | 1 [0 to 4] | 1 [0 to 3]
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 1-month post hospitalization for anxiety score; Test type: Superiority; p = 0.29, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.14 to 1.80] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 3-months post hospitalization for anxiety score; Test type: Superiority; p = 0.57, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.18 to 2.60] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 1-month post hospitalization for depression score; Test type: Superiority; p = 0.12, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 0.36, 95% CI 2-sided [0.10 to 1.30] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 3-months post hospitalization for depression score; Test type: Superiority; p = 0.48, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 0.62, 95% CI 2-sided [0.16 to 2.40] — [estimate comment as in outcome 5, analysis 1]

10. Secondary Outcome: Mental Health - Post-Traumatic Distress Using Impact of Events Scale-Revised (IES-R)
Description: The Impact of Events Scale-Revised (IES-R) is a self-reported questionnaire that measures the distress caused by traumatic events. Subjects respond to 22 questions using a 5-point scale ranging from 0 (not at all) to 4 (extremely). Total scores range from 0 to 88, with a higher score indicting the likely presence of post-traumatic stress disorder (PTSD).
Time Frame: 1 and 3-months post-hospitalization
Population: as for outcome 9
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 45 | 42
score on a scale
  1 month post hospitalization | 1 [0 to 9] | 3 [0 to 11]
  3 months post hospitalization: number analyzed (Participants) | 41 | 41
  3 months post hospitalization | 0 [0 to 0] | 0 [0 to 4]
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 1-month post hospitalization; Test type: Superiority; p = 0.56, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.39 to 5.60] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 3-months post hospitalization; Test type: Superiority; p = 0.02, proportional odds; proportional odds models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 9.16, 95% CI 2-sided [1.40 to 59.9] — [estimate comment as in outcome 5, analysis 1]

11. Secondary Outcome: Number of Participants With Allogeneic Red Blood Cell Transfusions
Description: Number (percentage) of patients transfused with allogeneic red blood cells
Time Frame: 3-months post-hospitalization
Population: No data was collected or analyzed for 1 participant in the anemia treatment bundle arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 51 | 48
Participants | 6 | 1
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; Test type: Superiority; p = 0.09, Regression, Logistic; adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 0.16, 95% CI 2-sided [0.02 to 1.40] — [estimate comment as in outcome 5, analysis 1]

12. Secondary Outcome: Number of Transfused Units of Allogeneic Red Blood Cells
Description: Number of transfused units from hospital discharge through 3-months post-hospitalization
Time Frame: 3 months post hospitalization
Population: No data was collected or analyzed for 1 participant in the anemia treatment bundle arm.
Measure: Median (Inter-Quartile Range); unit: Transfused units
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 51 | 48
Transfused units | 0 [0 to 0] | 0 [0 to 0]

13. Secondary Outcome: Unplanned Hospital Readmissions
Description: Number of subjects to experience an unplanned hospital readmission
Time Frame: 3 months and 12-months post-hospitalization
Population: No data was collected or analyzed for 1 participant in the anemia treatment bundle arm at 3-months post hospitalization. No data was collected or analyzed for 1 participant in the anemia treatment bundle arm at 12-months post hospitalization.
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 51 | 48
Participants
  3 months post hospitalization | 16 | 12
  12 months post hospitalization | 30 | 24
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 3-months post hospitalization; Test type: Superiority; p = 0.48, Regression, Logistic; logistic models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.30 to 1.80] — Estimates are odds ratios and correspond to the multiplicative increase in odds for the given event associated with intervention associated with active intervention

14. Secondary Outcome: Mortality
Description: Mortality from any cause
Time Frame: 3 months and 12-months post-hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 51 | 49
Participants
  3 months post hospitalization | 1 | 2
  12 months post hospitalization | 2 | 3
Statistical Analysis 1: Comparison: Control (Standard of Care) Group vs Anemia Treatment Bundle; 3-months post hospitalization; Test type: Superiority; p = 0.54, Regression, Logistic; logistic models adjusting for baseline hemoglobin, age, sex, and surgical vs. non-surgical admission; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.19 to 24.0] — [estimate comment as in outcome 13, analysis 1]

15. Secondary Outcome: Adverse Events Post-enrollment
Description: Venous thromboembolism, bloodstream infection, myocardial infarction, stroke
Time Frame: Hospital discharge (approximately 1 month), 3-months post-hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 51 | 49
Participants
  Venous Thromboembolism | 4 | 2
  Bloodstream Infection | 2 | 0
  Myocardial Infarction | 2 | 1
  Stroke | 0 | 2

16. Secondary Outcome: Accelerometry-measured Number of Steps Taken Per Day
Description: Home-based activity monitor daily step counts (optional, exploratory study component)
Time Frame: 1 and 3-months post-hospitalization
Population: No data was collected or analyzed for 33 participants in the control standard of care arm and 27 participants in the anemia treatment bundle arm.
Measure: Median (Full Range); unit: Number of steps per day
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 18 | 22
Number of steps per day
  1 month post hospitalization | 6481 [2690 to 14772] | 6017 [3046 to 9010]
  3 month post hospitalization | 8281 [2535 to 13816] | 6874 [2275 to 11972]

17. Secondary Outcome: Accelerometry-measured Daily Maximum Step Cadence
Description: Actigraphy evaluated daily Max Step Cadence - i.e., steps per minute (optional, exploratory study endpoint)
Time Frame: 1 month and 3 month post hospitalization
Population: as for outcome 16
Measure: Median (Full Range); unit: Steps per Minute
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
Number analyzed (Participants) | 18 | 22
Steps per Minute
  1 month post hospitalization | 67.0 [27.0 to 102.5] | 64.4 [29.8 to 109.5]
  3 months post hospitalization | 71.1 [34.3 to 106.3] | 61.4 [29.5 to 110.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline through approximately 3-months after hospitalization.
Description: Death was collected through 12 months post hospitalization; all other adverse events were collected from baseline through approximately 3-months post hospitalization.
Arm/Group | Control (Standard of Care) Group | Anemia Treatment Bundle
All-Cause Mortality (participants affected / at risk) | 2/51 | 3/49
Serious Adverse Events (participants affected / at risk) | 3/51 | 1/49
Other Adverse Events (participants affected / at risk) | 5/51 | 4/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Standard of Care) Group (N=51) | Anemia Treatment Bundle (N=49)
Bloodstream Infection (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Venous Thromboembolism (Vascular disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Standard of Care) Group (N=51) | Anemia Treatment Bundle (N=49)
Venous thromboembolism (Vascular disorders) | 4 (4) | 2 (2)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 1 (1)
Stroke (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT05167734/Prot_SAP_001.pdf
  • Informed Consent Form (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/34/NCT05167734/ICF_000.pdf